CLINICAL TRIAL: NCT04178837
Title: Role of Ultrasound Imaging in Diagnosis of Juvenile Idiopathic Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam eldeen Esmael Zayan, asmaa mohammed abd elhameed ali (amaeali), Assiut University
Other Study IDs: Us in JIA
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Juvenile idiopathic arthritis (JIA) is the most common chronic rheumatic disease of childhood and an important cause of acquired disability in children . Despite the heterogeneity, all forms of JIA are characterized by prolonged synovial inflammation that can cause cartilage and bone damage, with severe impairment of physical function and impact on the quality of life. The presence of joint involvement in JIA may be expressed by ultrasonography findings such as synovial proliferation, effusion, cartilage thinning and bone erosions. US has demonstrated higher sensitivity in detecting synovitis compared to clinical examination MSUS is commonly regarded as a very useful tool in children, as outlined by the results of recent national and international surveys among pediatric rheumatologists .For most of the respondents, MSUS owned particular relevance for the ability to detect subclinical synovitis and to improve the classification of patients in JIA subtypes, as guidance to intraarticular corticosteroid injections and for capturing early articular damage. In addition, some specific joints were considered as most suited to be studied by MSUS, specifically the midfoot, the ankle, the hip, the wrist, the small joints of hands and feet. .

DETAILED DESCRIPTION:
Juvenile idiopathic arthritis (JIA) is the most common chronic rheumatic disease of childhood and an important cause of acquired disability in children . Despite the heterogeneity, all forms of JIA are characterized by prolonged synovial inflammation that can cause cartilage and bone damage, with severe impairment of physical function and impact on the quality of life. The presence of joint involvement in JIA may be expressed by ultrasonography findings such as synovial proliferation, effusion, cartilage thinning and bone erosions. US has demonstrated higher sensitivity in detecting synovitis compared to clinical examination MSUS is commonly regarded as a very useful tool in children, as outlined by the results of recent national and international surveys among pediatric rheumatologists .For most of the respondents, MSUS owned particular relevance for the ability to detect subclinical synovitis and to improve the classification of patients in JIA subtypes, as guidance to intraarticular corticosteroid injections and for capturing early articular damage. In addition, some specific joints were considered as most suited to be studied by MSUS, specifically the midfoot, the ankle, the hip, the wrist, the small joints of hands and feet. .

ELIGIBILITY:
Inclusion Criteria:

* Age between 1-17 years only.
* Both sexes.
* children with any type of Juvenile Idiopathic Arthritis

  -Exclusion criteria
* Age above 17years.
* Children with arthritis of known cause.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children with any type of Juvenile Idiopathic Arthritis
Sampling Method: Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2020-02-24 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Role of Ultrasound imaging in diagnosis of juvenile idiopathic arthritis | 2019_2021
  Role of Ultrasound imaging in diagnosis activity &exacepation of juvenile idiopathic arthritis